CLINICAL TRIAL: NCT05236504
Title: Effects of a Novel Melatonin and Magnesium-Containing Pod on Sleep, Metabolism, Body Composition and Performance
Brief Title: Effects of a Novel Supplement on Sleep, Metabolism, Body Composition and Performance
Acronym: 4BETTSLEEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bettery S.A. (Industry)
Responsible Party: Principal Investigator, Filipe Teixeira, Innovation Manager, Bettery S.A.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Bettery LifeLab4BS
Record Dates: First submitted 2022-01-18; First posted 2022-02-11 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Sleep Hygiene; Sleep Disturbance
Keywords: Melatonin; Magnesium; Supplementation; Sleep; Resting metabolic rate; Body composition; Handgrip Strength
MeSH Terms: conditions — Sleep Hygiene; Parasomnias | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplement (Experimental): Melatonin and magnesium-containing pod
  Interventions: Dietary Supplement: Melatonin and magnesium-containing pod
- Placebo (Placebo Comparator): Placebo pod
  Interventions: Other: Placebo comparator

INTERVENTIONS:
Dietary Supplement: Melatonin and magnesium-containing pod — A 50-100mL hot water drink, obtained from a coffee pod machine, containing 1.9mg of melatonin and 200mg of magnesium in a powdered form, will be ingested 30 minutes before bedtime. Total duration of this intervention: 4 weeks, after which 1 week of washout will occur, before switching to the other intervention.
  Arms: Supplement
Other: Placebo comparator — A 50-100mL hot water drink of identical taste, obtained from an identical pod with the same ingredients except melatonin and magnesium, will be ingested 30 minutes before bedtime. Total duration of this intervention: 4 weeks, after which 1 week of washout will occur, before switching to the other intervention.
  Arms: Placebo

SUMMARY:
This study aimed to investigate the effects of a novel dietary supplement, consisting of melatonin and magnesium in a pod (coffee machine capsule) format, on sleep quality, stress, mood, sleepiness, biological rhythms, metabolism, body composition and performance, in individuals with sleep disturbances according with the Pittsburgh Sleep Quality Index. A randomized, double-blind, crossover trial will be conducted to compare the effects of the melatonin and magnesium-containing supplement against a placebo. The protocol comprises 4 weeks of supplementation with an experimental or placebo condition, with a week-long washout period. Biochemical markers of sleep and stress, actigraphy for sleep patterns and sleep hygiene, resting metabolic rate, food and fluid intake, body composition, and handgrip strength measures will be evaluated at baseline and 4 weeks post each randomly assigned intervention. The working hypothesis is that this innovative supplement will provide greater objective and subjective improvements regarding sleep patterns and quality, overall mood, biochemical markers of stress, resting metabolic rate, energy intake, body composition and strength, than the placebo comparator, due to the synergic effects of melatonin and magnesium.

DETAILED DESCRIPTION:
A randomized, double-blind, crossover design will be used to investigate the efficacy of a novel developed melatonin and magnesium supplement in pod (coffee machine capsule) format on sleep patterns and sleep quality, mood, sleepiness, biological rhythms, stress, metabolism, body composition and strength performance. Prior to the intervention, participants will be screened for inclusion and exclusion criteria, namely presenting with sleep disturbs according to Pittsburgh Sleep Quality Index (score >5), not working in shifts, not experiencing jet lag frequently (e.g., flight personnel), nor taking medication which could interfere with sleep. A total of 35 individuals suffering from sleep disturbs will engage in 4 weeks of supplementation with melatonin and magnesium or placebo, separated by 1 week of washout, after which the second experimental condition will be conducted (4 weeks placebo or supplementation with melatonin and magnesium). At baseline and 4 weeks post each, randomly assigned intervention, participants will experience measurements of resting metabolic rate, body composition and strength, as well as the collection of saliva to measure melatonin and cortisol. Validated questionnaires on sleep quality, mood, sleepiness, and biological rhythms will also be applied and nutritional intake will be quantified and assessed for frequency and timing on the three occasions. Throughout the 8 weeks of supplementation, participants will use an actigraphy device continuously to evaluate sleep and awaken motor activity, and compliance to the assigned intervention will be confirmed in each visit to the laboratories.

In order to achieve the main goal of the study, assessments will take place in the morning (starting at 7:00 a.m.), after an overnight fast. Wearing minimal clothing and no shoes, participants will be weighed on a scale and have their height measured on a stadiometer (Seca, Hamburg, Germany). Body composition, namely bone mineral content, fat mass and fat free mass, will be assessed by dual energy X-ray absorptiometry (DXA) (Horizon Wi, Hologic, Waltham, USA). Total body water and its intra and extracellular compartments will be estimated from whole body resistance (R) and reactance (Xc), measured through bioelectrical impedance analysis (BIA), using a single frequency device of 50 kHz (BIA-101, RJL/Akern Systems, Firenze, Italy). From the raw R and Xc data, the phase angle will additionally be determined, using the Akern Software.

Resting metabolic rate (RMR) will be measured by indirect calorimetry, using a canopy ventilated open-circuit system (Quark, Cosmed, Italy). Participants will arrive to the laboratory in an overnight-fasted state, having refrained from exercise, caffeine, and alcohol consumption in the 12h before assessments. The equipment will be calibrated daily according to standard procedures. Participants will rest in supine position prior to the start of the measurement. Data will be collected for ≥15min with the first 5min being dismissed, according to protocol. The average resting metabolic rate will be considered the period of 5min of the test with lower coefficient of variance.

The handgrip strength test will be used to evaluate the maximal isometric force of the muscles of the hand and forearm. Using a portable hand dynamometer (JAMAR, Sammons Preston, Bolingbrook, IL, USA), participants will be tested for both hands alternately, in a stand-up position. The maximal force generated out of 3 attempts will be considered for analysis.

For biochemical markers, saliva will be collected in salivettes. Saliva will be used to measure melatonin and cortisol using Enzyme-Linked Immunosorbent Assay (ELISA).

In an interview with a Registered Dietitian on the three visits to the labs, participants will report food and fluid intake in the 24h before. Timing of the meals, cooking/preparation methods, product specificities and estimated portion sizes will be recorded. To support this methodology, a validated food frequency questionnaire will be applied to assess for type and frequency of food and drink consumption, during the month-long interventions. Together, these data will allow to identify the pattern of ingestion (quantity, quality and timing) of key foods (i.e. kiwifruit, tart cherry, milk, valerian tea) and nutrients (i.e. total energy intake (TEI), total carbohydrate (CHO) in grams and as a %TEI, high glycaemic index CHO, low glycaemic index CHO, tryptophan, caffeine, alcohol) with potential impact on sleep parameters. Dietary intake will be quantified using a dietary analysis software (Nutritics Research Edition (v5.09), Dublin, Ireland). Participants will be instructed to maintain their eating habits throughout the 9 weeks of the investigation.

At baseline and after both interventions, subjects will be asked to fill in the Portuguese validated questionnaires: Pittsburgh Sleep Quality Index (PSQI), Profile of Mood States (POMS), Epworth Sleepiness Scale (ESS) and Horne & Oestberg Morningness-Eveningness Questionnaire (MEQ), to evaluate subjective sleep quality, mood, sleepiness, and biological rhythms, respectively.

In order to objectively evaluate sleep parameters (i.e., sleep latency, total sleep time, sleep efficiency) during the night and motor activity during the day, as well as to quantify total energy expenditure and activity energy expenditure throughout the 8 weeks of supplementation, participants will be asked to wear an activity monitor device with a validated 3-axis accelerometer (ActiGraph GT9X Link, Florida, USA) continuously, during the day and at night.

Randomization and Supplementation: The order of the interventions (treatment or placebo) will be randomized by an external investigator. All eligible participants will be assigned to the same group initially, but will experience both conditions in a crossover manner. The investigator responsible for the sample randomization and the distribution of the supplements is not directly involved in participants' eligibility interview nor in data collection.

Sample justification and sample size: According to a recent systematic review and meta-analysis of randomized controlled trials (PMID: 33417003), melatonin levels decrease with age, while the incidence of sleep disturbances increases proportionally. However, a decline in melatonin levels is not typically observed before the age of 35, while after the age of 55, other comorbidities and/or the intake of medication may instead explain alterations to the sleep cycle. Notwithstanding, a cohort study looking at a large spectrum of ages (PMID: 21091391) has demonstrated the short- and long-term efficacy of 2mg of prolonged-release melatonin in insomnia patients between 18-80 years old, particularly those aged 55 and over. Considering the similar dosage to that of this novel formula (1.9mg of melatonin), recruiting a sample of participants between the ages of 35-55 is one of the inclusion criteria. People who work in shifts or who may experience jet lag due to their profession (e.g., flight personnel) are excluded on the basis that irregular sleep patterns may interfere with sleep quality. Considering the literature presented, the investigators have decided to establish a similar sample size and study duration (4 weeks + 4 weeks) to that of previous studies. Sample size was calculated using g power version 3.1., based on an effect size of 0.25, power of 0.8 and alpha 0.05. A sample of 28 subjects was deemed required. Assuming a dropout of 25%, the researchers have pursued a sample of 35 participants.

Statistics: All statistical analyses will be carried out using IBM SPSS Statistics (NY, IBM). Basic descriptive data will be used to characterize the participants in the study and all variables will be checked for normality, using Shapiro-Wilk test. All participants will initially be assigned to the same intervention group. Time and time-by-group interactions will be evaluated by Mixed ANOVA. The equality of the matrix of variance and sphericity will be explored with the Levene F test and Mauchly's test, respectively. Overall significance level for α will be set at p ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Pittsburgh Sleep Quality Index >5 as an indicator of sleep disturbance.

Exclusion Criteria:

* Taking medication which interferes with sleep;
* Shift workers;
* Workers who may experience jet lag (e.g. flight personnel).

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-11-28 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Biochemical sleep marker - Change in salivary melatonin | Baseline, week 4 (post-intervention 1) and week 9 (post-intervention 2)
  Salivary melatonin (pg/mL) will be assessed by enzyme-linked immunosorbent assay (ELISA)
Biochemical stress marker - Change in salivary cortisol | Baseline, week 4 (post-intervention 1) and week 9 (post-intervention 2)
  Salivary cortisol (ug/dL) will be assessed by ELISA
Sleep parameter - Change in sleep latency | Daily throughout the 4 weeks of intervention 1 and 4 weeks of intervention 2
  Sleep latency (minutes) will be assessed by actigraphy
Sleep parameter - Change in total sleep time | Baseline, week 4 (post-intervention 1) and week 9 (post-intervention 2)
  Total sleep time (hours) will be assessed by actigraphy
Sleep parameter - Change in sleep efficiency | Baseline, week 4 (post-intervention 1) and week 9 (post-intervention 2)
  Sleep efficiency (percent) will be assessed by actigraphy
Sleep parameter - Change in sleep quality | Baseline, week 4 (post-intervention 1) and week 9 (post-intervention 2)
  Change in sleep quality (Pittsburgh Sleep Quality Index (PSQI) score) will be assessed by the validated Portuguese version of the PSQI. The PSQI global score, results from the sum of 7 component scores (0-3) and has a possible range of 0-21 points. A global PSQI score ≤ 5 identifies a good sleeper and >5 a poor sleeper.
Sleep parameter - Change in mood states | Baseline, week 4 (post-intervention 1) and week 9 (post-intervention 2)
  Change in mood states ('Profile of Mood States' (POMS) score) will be assessed by the validated Portuguese adaptation (Viana, Almeida and Santos, 2001) of a short version of the POMS. A total mood disturbance score is calculated by summing the totals for the 5 negative subscales (tension, depression, fatigue, confusion, anger) and subtracting the positive subscale (vigour), adding 100 to avoid a negative global result. Scores for each item are recorded as 0 for 'not at all' up to 4 for 'extremely'. Total mood disturbance scores can range between -64 and 100. Higher scores indicate a greater degree of mood disturbance.
Sleep parameter - Change in daytime sleepiness | Baseline, week 4 (post-intervention 1) and week 9 (post-intervention 2)
  Daytime sleepiness (Epworth Sleepiness Scale (ESS) score) will be assessed by the validated Portuguese version (CEISUC, 2001) of the questionnaire. ESS global score results from the sum of 8 item scores (0-3) and can range from 0 to 24 points. The higher the ESS score, the higher that person's average sleep propensity in daily life: 0-5 Lower Normal Daytime Sleepiness; 6-10 Higher Normal Daytime Sleepiness; 11-12 Mild Excessive Daytime Sleepiness; 13-15 Moderate Excessive Daytime Sleepiness; 16-24 Severe Excessive Daytime Sleepiness.
Sleep parameter - Change in biological rhythms | Baseline, week 4 (post-intervention 1) and week 9 (post-intervention 2)
  Change in biological rhythms ('Morningness-Eveningness Questionnaire' (MEQ) score) will be assessed by the validated Portuguese version (Silvério, Silva and Macedo, 1998) of the MEQ. Four sections of the 16-item scale are assigned a value of 1 through 5, while the remaining twelve questions are assigned a value of 1 through 4. To obtain a global score, the sum of the components is converted to a 5-point scale: definitely morning type (>59); moderately morning type (54-59); neither type (43-53); moderately evening type (31-42); and definitely evening type (<31). Morningness-eveningness scores can range between 16-68.
Metabolic parameter - Change in resting metabolic rate (RMR) | Baseline, week 4 (post-intervention 1) and week 9 (post-intervention 2)
  RMR (kcal) will be assessed by indirect calorimetry
Dietary intake parameter - Change in total energy intake (TEI) | Baseline, week 4 (post-intervention 1) and week 9 (post-intervention 2)
  TEI (kcal/day) will be assessed by 24h recall and quantified using a dietary analysis software
Dietary intake parameter - Change in total carbohydrate (CHO) intake | Baseline, week 4 (post-intervention 1) and week 9 (post-intervention 2)
  CHO intake (g/day; percent of TEI) will be assessed by 24h recall and quantified using a dietary analysis software
Dietary intake parameter - Change in high and low glycemic index CHO | Baseline, week 4 (post-intervention 1) and week 9 (post-intervention 2)
  High and low glycemic index CHO (g/day) will be assessed by 24h recall and quantified using a dietary analysis software
Dietary intake parameter - Change in triptophan intake | Baseline, week 4 (post-intervention 1) and week 9 (post-intervention 2)
  Triptophan intake (g/day) will be assessed by 24h recall and quantified using a dietary analysis software
Dietary intake parameter - Change in caffeine intake | Baseline, week 4 (post-intervention 1) and week 9 (post-intervention 2)
  Caffeine intake (mg/day) will be assessed by 24h recall and quantified using a dietary analysis software
Dietary intake parameter - Change in alcohol intake | Baseline, week 4 (post-intervention 1) and week 9 (post-intervention 2)
  Alcohol intake (g/day) will be assessed by 24h recall and quantified using a dietary analysis software
Dietary intake parameter - Change in the timing of dietary intake | Baseline, week 4 (post-intervention 1) and week 9 (post-intervention 2)
  Timing of dietary intake (hours) will be assessed for each food and drink mentioned in the 24h recall
Dietary intake parameter - Change in the frequency of dietary intake | Baseline, week 4 (post-intervention 1) and week 9 (post-intervention 2)
  Frequency of dietary intake (days/week or days/month) will be assessed using a validated food frequency questionnaire

SECONDARY OUTCOMES:
Dietary intake parameter - Change in protein intake | Baseline, week 4 (post-intervention 1) and week 9 (post-intervention 2)
  Protein intake (g/day) will be assessed by 24h recall and quantified using a dietary analysis software
Dietary intake parameter - Change in fat intake | Baseline, week 4 (post-intervention 1) and week 9 (post-intervention 2)
  Fat intake (g/day) will be assessed by 24h recall and quantified using a dietary analysis software
Body composition parameter - Change in fat free mass (FFM) | Baseline, week 4 (post-intervention 1) and week 9 (post-intervention 2)
  FFM (kg) will be assessed by dual energy X-ray absorptiometry
Body composition parameter - Change in fat mass (FM) | Baseline, week 4 (post-intervention 1) and week 9 (post-intervention 2)
  FM (percent) will be assessed by dual energy X-ray absorptiometry
Body composition parameter - Change in visceral adipose tissue (VAT) | Baseline, week 4 (post-intervention 1) and week 9 (post-intervention 2)
  VAT Area (cm^2) will be assessed by dual energy X-ray absorptiometry
Body composition parameter - Change in body water | Baseline, week 4 (post-intervention 1) and week 9 (post-intervention 2)
  Total body water, intracellular water and extracellular water (L) will be assessed by bioelectrical impedance analysis
Body composition parameter - Change in phase angle | Baseline, week 4 (post-intervention 1) and week 9 (post-intervention 2)
  Phase angle (degree) will be assessed by bioelectrical impedance analysis
Performance parameter - Change in strength | Baseline, week 4 (post-intervention 1) and week 9 (post-intervention 2)
  Maximal isometric forearm strength (N) will be assessed using a handgrip dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- Bettery, S.A., Porto Salvo, Oeiras, Portugal

IPD SHARING:
Plan to Share IPD: No